CLINICAL TRIAL: NCT04867343
Title: Pharmacokinetics, Safety and Efficacy of HR020602 Injection in Children Undergoing General Anesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR020602-201
Record Dates: First submitted 2021-04-24; First posted 2021-04-30 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Used to Induce and Implement General Anesthesia in Combination With Sedative Anesthetics (Such as Propofol)

STUDY DESIGN:
Intervention Model Description: This study is divided into two stages: the first stage is a dose verification trial, with a multicenter, open, single arm trial design, which is planned to enroll 10 children with general anesthesia surgery (all using HR020602 injection); If the result shows that the dose is low, 10 children under general anesthesia will be included again for higher dose verification. The second stage is designed as a multicenter, randomized, double-blind, parallel control trial with positive drugs, which is planned to include 25 children with general anesthesia surgery in the test group and 25 children in the control group. There should be at least 20 patients in each of [2,12] and [12,18）age groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HR020602 injection (Experimental)
  Interventions: Drug: HR020602 injection
- fentanyl injection + remifentanil injection (Active Comparator)
  Interventions: Drug: fentanyl injection ； remifentanil injection

INTERVENTIONS:
Drug: HR020602 injection — HR020602 injection
  Arms: HR020602 injection
Drug: fentanyl injection ； remifentanil injection — fentanyl injection + remifentanil injection
  Arms: fentanyl injection + remifentanil injection

SUMMARY:
This study is divided into two stages: the first stage is a dose verification trial, with a multicenter, open, single arm trial design, which is planned to enroll 10 children with general anesthesia surgery (all using HR020602 injection); If the result shows that the dose is low, 10 children under general anesthesia will be included again for higher dose verification.The second stage is designed as a multicenter, randomized, double-blind, parallel control trial with positive drugs, which is planned to include 25 children with general anesthesia surgery in the test group and 25 children in the control group. There should be at least 20 patients in each of [2,12] and [12,18）age groups.

ELIGIBILITY:
Inclusion Criteria:

1. 2 years old ≤age<18 years old, regardless of gender;
2. General anesthesia is planned;
3. ASA score grade I ~ II; 4）Able to sign the informed consent.

Exclusion Criteria:

1. Children with general anesthesia contraindications;
2. With diseases that are not suitable for the study in the scheme;
3. Abnormal liver and kidney function in screening stage;
4. Abnormal coagulation function;
5. Serum electrolyte abnormality;
6. Subjects intolerant or allergic to the study drugs;
7. Recently received other narcotic drugs or other drugs that affect the metabolism of study drugs;
8. The child thought to be unsuitable for the study, as determined by the investigator.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
The success rate of anesthesia induction | Within 5 minutesafter propofol medium /long chain fat emulsion administration

SECONDARY OUTCOMES:
The success rate of anesthesia maintenance | Procedure (During the period from the beginning of anesthesia maintenance drugs to the end of anesthesia)
Anesthesia recovery time | The time from stopping using anesthetic drugs (propofol medium/long-chain fat emulsion) to the time when the subject wakes up (opening eyes as instructed)
The dosage of propofol medium/long chain fat emulsion during anesthesia maintenance period | Procedure (During the period from the beginning of anesthesia maintenance drugs to the end of anesthesia)
The dosage of opioids during anesthesia maintenance period | Procedure (During the period from the beginning of anesthesia maintenance drugs to the end of anesthesia)
Clearance rate (CL), apparent volume of distribution (V) and inter individual variation (CV%) of parameters | PK blood collection are to be performed at 5 time points during Day 1-Day 2)
The incidence and severity of adverse events during the trial | Through study completion, about 3-10 days)
The incidence of adverse reactions of the mental system | Within 1 hour after awakening)
Proportion of subjects with unstable hemodynamics (blood pressure, heart rate) | Through study completion, about 3-10 days)

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital, Tianjin Medical University, Tianjin, Tianjin Municipality, China